CLINICAL TRIAL: NCT00784108
Title: Non-contact Imaging Device (Camera) Can Help Improve Treatment for Patients With Basal Cell Carcinoma.
Brief Title: Optimizing Photodynamic Therapy of Cutaneous Neoplastic Diseases Via Structured Illumination and Real-time Dosimetry.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D., Professor Departments of Dermatology and Surgery, University of California, Irvine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20086439
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Skin Cancer; Signs and Symptoms
MeSH Terms: conditions — Skin Neoplasms; Signs and Symptoms | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diagnostic tool (Other): Modulated Imaging measure effect of Photodynamic therapy treatment
  Interventions: Device: Modulated Imaging (MI)
- Photodynamic therapy (Other): Modulated Imaging measure effect of Photodynamic therapy treatment
  Interventions: Other: Photodynamic therapy

INTERVENTIONS:
Device: Modulated Imaging (MI) — Modulated Imaging measure effect of Photodynamic therapy treatment
  Other Names: non-contact optical imaging device (camera)
  Arms: Diagnostic tool
Other: Photodynamic therapy — Modulated Imaging measure effect of Photodynamic therapy treatment
  Arms: Photodynamic therapy

SUMMARY:
The purpose of this study is to evaluate native tissue optical properties and photosensitizer optical properties in vivo with a novel, non-contact optical imaging device call Modulated Imaging to help optimize the laser exposure in future photodynamic treatment for patients with skin cancer.

Photodynamic therapy involves the administration of a tumor-localizing photosensitizing agent that, when illuminated with the proper wavelength of light, can result in photochemical processes that cause irreversible damage to tumor tissues. Photodynamic therapy is non-invasive and has been shown to be effective in the treatment of skin cancer while producing excellent aesthetic appearance and psychological well-being in patients that normally would require invasive excisions.

DETAILED DESCRIPTION:
The current standard of care for skin cancer is excision, curettage and electrodesiccation and/or cryosurgery.

The Modulated Imaging can measure tissue optical properties that effect the Photodynamic therapy treatment process can show spectral absorption and scattering coefficients, oxy- and deoxy-hemoglobin, water, melanin and use that information to provide customized laser light treatment.

The researchers can use an imaging system that can characterize the tissue and photosensitizer optical properties and use that information to drive a treatment light projection system that can spatially optimize the light irradiance for personalized treatment, thus improving outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Biopsy proven diagnosis of a basal cell carcinoma in a non-facial area

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Breast feeding.
* photosensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Measure tissue optical properties | 4 weeks
  Modulated Imaging measure effect of Photodynamic therapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Kelly, MD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States